CLINICAL TRIAL: NCT05469399
Title: The Effect of Game-Based Virtual Reality Learning Method on the Learning Outcomes of Nursing Students for Postoperative Admission of the Patient to the Clinic
Brief Title: Admission of the Patient to the Clinic After Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Burcu Opak Yücel, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BOYucel
Record Dates: First submitted 2022-06-09; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Post Operative Pain; Post-Op Hemorrhage; Postoperative Hypothermia; Nurse's Role
Keywords: post operative pain; post operative hemorrhage; nursing care
MeSH Terms: conditions — Pain, Postoperative; Postoperative Hemorrhage | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GBVRLPCA (Experimental): Students in the experimental group will be given a knowledge test, an objectively structured clinical exam for skill assessment, theoretical lectures, and a game practice for a week. One week later, students will be given a knowledge test, an objectively structured clinical exam for skill evaluation, and an evaluation form for game practice.
  Interventions: Other: Experimental Group
- Control Group (Active Comparator): The students in the control group will be given a knowledge test, an objectively structured clinical exam for skill assessment, theoretical lessons, and no application will be made for a week. After one week, students will be given a knowledge test and an objective structured clinical exam for skill assessment.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Experimental Group — Students will be given a "knowledge test" and an "objective structured clinical exam for skill assessment" (Initial knowledge and skill assessment). After these applications, the students will be given a theoretical course on the admission of the patient to the clinic after the operation. After the theoretical lesson, a link for the virtual reality game application consisting of three different cases will be sent to the students for them to play on the phone and computer. Students will play this game application for a week. After the game application process, students will be given a "knowledge test", an "objective structured clinical exam for skill assessment" (final knowledge and skill assessment).
  Arms: GBVRLPCA
Other: Control Group — Students will be given a "knowledge test" and an "objective structured clinical exam for skill assessment" (Initial knowledge and skill assessment). No application will be made to the students for one week. One week later, students will be given a "knowledge test", an "objective structured clinical exam for skill assessment" (final knowledge and skill assessment).
  Arms: Control Group

SUMMARY:
Aim:This research was designed as a randomized controlled study to examine the effect of the game-based virtual reality learning method on the patient's post-operative admission to the clinic on the learning outcomes of the students.

Desing: This study was designed as a randomized controlled study to examine the effect of the game-based virtual reality learning method on the patient's post-operative admission to the clinic on the learning outcomes of the students.

Metod: The universe of the research will be nursing students who have taken the Surgical Diseases Nursing Course at Gazi University Faculty of Health Sciences Nursing Department in the 2021-2022 academic year. As a result of the power analysis using the G-power 3.1.9.7 package program; The effect size was calculated as 0.40 (It was seen from the literature studies that the effect size of the change in the knowledge score of the two groups was large effect size), and the total number of 68 samples is sufficient with 90% power, 5% margin of error, 95% confidence level, 20% drop-out Considering the rate of study, it was found sufficient to work with at least 82 people (Experiment: 41, Control: 41). For research data, "descriptive features form", "knowledge test form", "skill evaluation checklist", "student opinions form about game-based virtual reality game application", egameflow scale will be used.

ELIGIBILITY:
Inclusion Criteria:

* Students who voluntarily participated in the study
* Students who have taken all the subjects of the Surgical Diseases Nursing Course
* Students with smartphones, tablets, computers
* Students with internet access

Exclusion Criteria:

* Students who do not participate in the theoretical training
* Students who take the Surgical Diseases Nursing Course from below
* Students who do not want to continue the research
* Students who do not fill out the data collection forms at any stage
* Students who do not participate in the virtual reality-based game application
* Students who do not participate in any of the skills assessment
* Students who fill in the data collection forms incompletely

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
skills assessment | change in skill assessment for one week
  objective structured clinical exam
knowledge level | change in skill assessment for one week
  knowledge test

IPD SHARING:
Plan to Share IPD: No